CLINICAL TRIAL: NCT06103942
Title: Automated Carbon Dioxide Angiography in Comparison to Iodinated Contrast Medium Angiography During Fenestrated/Branched Endovascular Abdominal Aortic Aneurysm Repair (F/B-EVAR)
Brief Title: Automated Carbon Dioxide Angiography in Fenestrated/Branched Endovascular Abdominal Aortic Aneurysm Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: Nov2023
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Thoracoabdominal Aortic Aneurysm
Keywords: FEVAR; BEVAR; CO2; complex aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CO2 angiography — A supplemental CO2 angiography will be performed before and after the stent graft placement.

SUMMARY:
Carbon Dioxide (CO2)-based angiography is a digital subtraction angiography (DSA), where CO2 is used as an intra-arterial contrast agent.

Now, with the availability of an automated CO2 injector system (Angiodroid Srl, Italy) and the improvement in image acquisition protocols, CO2 angiography is increasingly used for vascular imaging and endovascular procedures.

Fenestrated and branched endovascular aortic repair (F/B-EVAR) for thoracoabdominal aortic aneurysms (TAAAs) is nowadays considered the treatment of first choice, due to its reduced procedure-related morbidity and mortality, when compared to open repair.

A peculiarity of these procedures is the need of high volumes of contrast media, which are not needed in case of open repair. This increases the related risk of impaired kidney function at the short- and long-term.

The present study will specifically examine the safety of the use of CO2 as intra-arterial contrast agent using the Angiodroid automated CO2-injection system during F/B-EVAR procedures. Furthermore, the current study will focus on image quality during the different steps of the procedure with the aim of standardize injection parameters (volume and pressure) for the detection of the ostium of the visceral vessels as well as of the iliac arteries, all defined as target vessels.

DETAILED DESCRIPTION:
Carbon Dioxide (CO2)-based angiography is a digital subtraction angiography (DSA), where CO2 is used as an intra-arterial contrast agent. This practice started in 1970s and it is commonly used for patients who have an impaired renal function, allergy to iodinated contrast media (ICM) or that could have a contrast-induced nephropathy (CIN) risk.

Carbon dioxide is an effective and low-risk alternative to ICM, which is nowadays used in endovascular procedures, thanks to its unique properties, such as no risk for nephrotoxicity or allergic reaction. For many years, the two most important restrictions for this technique consisted of: 1) the absence of a delivery system that could minimize the risk of air contamination during the CO2 angiography and allow controlled injection (in terms of pressure and volume of injection) of the CO2 and 2) the absence of a customized imaging protocol for a better visualization of CO2 during DSA acquisition.

Now, with the availability of an automated CO2 injector system (Angiodroid Srl, Italy) and the improvement in image acquisition protocols, CO2 angiography is increasingly used for vascular imaging and endovascular procedures.

Fenestrated and branched endovascular aortic repair (F/B-EVAR) for thoracoabdominal aortic aneurysms (TAAAs) is nowadays considered the treatment of first choice, due to its reduced procedure-related morbidity and mortality, when compared to open repair.

A peculiarity of these procedures is the need of high volumes of contrast media, which are not needed in case of open repair. This increases the related risk of impaired kidney function at the short- and long-term.

The literature on CO2 angiography still lacks on studies regarding the systematic use of the technique in F/B-EVAR procedures.

The present study will specifically examine the safety of the use of CO2 as intra-arterial contrast agent using the Angiodroid automated CO2-injection system during F/B-EVAR procedures. Furthermore, the current study will focus on image quality during the different steps of the procedure with the aim of standardize injection parameters (volume and pressure) for the detection of the ostium of the visceral vessels as well as of the iliac arteries, all defined as target vessels.

The main study hypothesis is that the automated standardized injection of CO2 could provide the same angiographic information and image quality as ICM, which is nowadays used as standard contrast agent in endovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for treatment of complex TAAA according to accepted international guidelines
* Provided informed consent

Exclusion Criteria:

* Severe COPD (Chronic Obstructive Pulmonary Disease), GOLD Stage 3 and 4
* Known atrium- or ventricular septal defect with right-left-shunt
* Current participation in other interventional studies

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a formal indication to an endovascular treatment of complex throacoabdominal aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | at the time the intervention
  Technical success in terms of detecting the ostium of the visceral vessels as well as of the hypogastric arteries (defined as 100% accuracy when compared to the iodinated contrast agent angiography)
CO2 sensitivity and specificity compared to iodinated contrast agent angiography | at the time the intervention
  CO2 sensitivity and specificity compared to iodinated contrast agent angiography in detecting dissections, stenosis, occlusions or bleeding of the target vessel. The comparison will be blinded and retrospective.

SECONDARY OUTCOMES:
Image quality | at the time the intervention
  Image quality with regard to the CO2 angiography defined as poor, moderate and good. The analysis of the images will be retrospective.

OTHER OUTCOMES:
Safety endpoints | within the first postoperative 24 hours
  Any adverse event within the first postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Asciutto, MD, PhD, Principal Investigator — Uppsala University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rolland Y, Duvauferrier R, Lucas A, Gourlay C, Morcet N, Rambeau M, Chaperon J. Lower limb angiography: a prospective study comparing carbon dioxide with iodinated contrast material in 30 patients. AJR Am J Roentgenol. 1998 Aug;171(2):333-7. doi: 10.2214/ajr.171.2.9694446.
- [Result] Palena LM, Diaz-Sandoval LJ, Candeo A, Brigato C, Sultato E, Manzi M. Automated Carbon Dioxide Angiography for the Evaluation and Endovascular Treatment of Diabetic Patients With Critical Limb Ischemia. J Endovasc Ther. 2016 Feb;23(1):40-8. doi: 10.1177/1526602815616924. Epub 2015 Nov 13. PMID 26567126
- [Result] Scalise F, Novelli E, Auguadro C, Casali V, Manfredi M, Zannoli R. Automated carbon dioxide digital angiography for lower-limb arterial disease evaluation: safety assessment and comparison with standard iodinated contrast media angiography. J Invasive Cardiol. 2015 Jan;27(1):20-6. PMID 25589696
- [Result] Seeger JM, Self S, Harward TR, Flynn TC, Hawkins IF Jr. Carbon dioxide gas as an arterial contrast agent. Ann Surg. 1993 Jun;217(6):688-97; discussion 697-8. doi: 10.1097/00000658-199306000-00011. PMID 8507115
- [Result] Caridi JG, Hawkins IF Jr. CO2 digital subtraction angiography: potential complications and their prevention. J Vasc Interv Radiol. 1997 May-Jun;8(3):383-91. doi: 10.1016/s1051-0443(97)70577-3. No abstract available. PMID 9152911
- [Result] Bettmann MA, D'Agostino R, Juravsky LI, Jeffery RF, Tottle A, Goudey CP. Carbon dioxide as an angiographic contrast agent. A prospective randomized trial. Invest Radiol. 1994 Jun;29 Suppl 2:S45-6. doi: 10.1097/00004424-199406001-00016. No abstract available. PMID 7928269
- [Result] Hawkins IF Jr, Wilcox CS, Kerns SR, Sabatelli FW. CO2 digital angiography: a safer contrast agent for renal vascular imaging? Am J Kidney Dis. 1994 Oct;24(4):685-94. doi: 10.1016/s0272-6386(12)80232-0. PMID 7942829
- [Result] D'Oria M, Wanhainen A, Lindstrom D, Tegler G, Mani K. Editor's Choice - Pre-Operative Moderate to Severe Chronic Kidney Disease is Associated with Worse Short-Term and Mid-Term Outcomes in Patients Undergoing Fenestrated-Branched Endovascular Aortic Repair. Eur J Vasc Endovasc Surg. 2021 Dec;62(6):859-868. doi: 10.1016/j.ejvs.2021.08.033. Epub 2021 Oct 27. PMID 34716095
- [Result] Gallitto E, Faggioli G, Vacirca A, Pini R, Mascoli C, Fenelli C, Logiacco A, Abualhin M, Gargiulo M. The benefit of combined carbon dioxide automated angiography and fusion imaging in preserving perioperative renal function in fenestrated endografting. J Vasc Surg. 2020 Dec;72(6):1906-1916. doi: 10.1016/j.jvs.2020.02.051. Epub 2020 Apr 8. PMID 32276017
- [Result] Chisci E, Michelagnoli S, Masciello F, Turini F, Panci S, Troisi N. Benefits and Role of Carbon Dioxide Angiography in Case of Misalignment Between Fenestration and Target Vessel During Fenestrated Endovascular Aneurysm Repair. J Endovasc Ther. 2022 Feb;29(1):7-10. doi: 10.1177/15266028211032955. Epub 2021 Aug 8. PMID 34369173
- [Result] Geisbusch S, Kuehnl A, Salvermoser M, Reutersberg B, Trenner M, Eckstein HH. Editor's Choice - Hospital Incidence, Treatment, and In Hospital Mortality Following Open and Endovascular Surgery for Thoraco-abdominal Aortic Aneurysms in Germany from 2005 to 2014: Secondary Data Analysis of the Nationwide German DRG Microdata. Eur J Vasc Endovasc Surg. 2019 Apr;57(4):488-498. doi: 10.1016/j.ejvs.2018.10.030. Epub 2019 Feb 7. PMID 30745030
- [Result] de Lachomette MF, Della N, Maucort-Boulch D, Duprey A, Rosset E, Feugier P, Lermusiaux P, Albertini JN, Millon A. Renal Function after Fenestrated or Branched Endovascular Aortic Repair: The Early Impairment Predictive Factors. Ann Vasc Surg. 2017 Apr;40:1-9. doi: 10.1016/j.avsg.2016.06.014. Epub 2016 Aug 27. PMID 27575304